CLINICAL TRIAL: NCT01520220
Title: A Phase 1 Study of LY2784544 Testing Alternative Dosing Regimens in Patients With Myeloproliferative Neoplasms
Brief Title: Study of LY2784544 Testing Alternative Dosing in Participants With Myeloproliferative Neoplasms
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14539; I3X-MC-JHTC (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-01-10; First posted 2012-01-27 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Myeloproliferative Neoplasms of; Polycythemia Vera; Essential Thrombocythemia; Myelofibrosis
MeSH Terms: conditions — Polycythemia Vera; Thrombocythemia, Essential; Primary Myelofibrosis | interventions — LY2784544

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part A: LY2784544 Dosing Regimen A (Experimental): LY2784544 will be taken by mouth per a specified schedule. Different participants will be treated at different doses until reaching the highest dose a participant can tolerate. Each cycle is 28 days.
  Interventions: Drug: LY2784544
- Part A: LY2784544 Dosing Regimen B (Experimental): LY2784544 will be taken by mouth per a specified schedule. Different participants will be treated at different doses until reaching the highest dose a participant can tolerate. Each cycle is 28 days.
  Interventions: Drug: LY2784544
- Part B: LY2784544 Dosing Regimen A (Experimental): LY2784544 will be taken by mouth per a specified schedule. Different participants will be treated at different doses from Part A that are determined to be safe and have potential clinical merit. Each cycle is 28 days.
  Interventions: Drug: LY2784544
- Part B: LY2784544 Dosing Regimen B (Experimental): LY2784544 will be taken by mouth per a specified schedule. Different participants will be treated at different doses from Part A that are determined to be safe and have potential clinical merit. Each cycle is 28 days.
  Interventions: Drug: LY2784544

INTERVENTIONS:
Drug: LY2784544 — LY2784544 will be taken by mouth per a specified schedule. Each cycle is 28 days.

SUMMARY:
The purpose of this study is to determine a dose of LY2784544 that may be safely administered to participants with myeloproliferative neoplasms.

ELIGIBILITY:
Inclusion Criteria:

Have a diagnosis of polycythemia vera (PV), essential thrombocythemia (ET), or myelofibrosis (MF, primary or secondary) PV and ET participants must have failed or are intolerant of standard therapies or refuse to take standard medications

MF participants must meet at least one of the following criteria:

* Have intermediate-1, intermediate-2, or high-risk MF according to the Dynamic International Prognostic Scoring System (DIPSS) plus; or
* Have symptomatic MF with spleen greater than 10 cm below left costal margin; or
* Have post-polycythemic MF (post-PV MF); or
* Have post-essential thrombocythemic MF (post-ET MF)

All participants must meet the following criteria:

* Have given written informed consent prior to any study-specific procedures
* Have adequate organ function, including:
* Hepatic: Direct bilirubin less than or equal to 1.5 times upper limits of normal (ULN), alanine transaminase (ALT), and aspartate transaminase (AST) less than or equal to 2.5 times ULN
* Renal: Serum creatinine less than or equal to 1.5 times ULN
* Bone Marrow Reserve: Absolute neutrophil count (ANC) ≥1000/mcL, platelets ≥25,000/mcL, platelets ≥50,000 for PV or ET participants.
* Have a performance status of 0, 1, or 2 on the Eastern Cooperative Oncology Group (ECOG) scale
* Have discontinued all previous approved therapies for MF, including any chemotherapy, immunomodulating therapy (for example, thalidomide, interferon-alpha), immunosuppressive therapy (for example, corticosteroids >10 mg/day prednisone or equivalent), radiotherapy, and erythropoietin, thrombopoietin, or granulocyte colony-stimulating factor (GSF) for at least 14 days and recovered from the acute effects of therapy. Hydroxyurea used to control blood cell counts is permitted at study entry if the participant has been maintained on a stable dose for at least 4 weeks. Low dose acetylsalicylic acid (aspirin; 81 or 100 mg) is permitted as well
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Males and females with reproductive potential must agree to use medically approved contraceptive precautions during the study and for 3 months following the last dose of study drug
* Females with child-bearing potential must have had a negative urine pregnancy test less than or equal to 7 days before the first dose of study drug and must also not be breastfeeding
* Are able to swallow capsules/tablets
* For participants who have undergone recent major surgery, at least 28 days must have elapsed between surgery and study participation, and the participant must have achieved, in the opinion of the treating physician, at least a good recovery from the surgical procedure

Exclusion Criteria:

Potential participants may not be included in the study if any of the following apply during screening:

* Have received treatment within 14 days of the initial dose of study drug with an experimental agent that has not received regulatory approval for any indication
* Have a QTc interval >470 milliseconds (msec) using Bazett's formula
* Have serious preexisting medical conditions that, in the opinion of the investigator, would preclude participation in the study (for example, a gastrointestinal (GI) disorder causing clinically significant symptoms such as nausea, vomiting, and diarrhea, or malabsorption syndrome)
* Are currently being treated with agents that are metabolized by cytochrome P450 (CYP)3A4 with a narrow therapeutic margin (for example, alfentanil, cyclosporine,diergotamine, ergotamine, fentanyl, pimozide, quinidine, sirolimus, and tacrolimus) or CYP2B6 (for example, cyclophosphamide, ifosfamide, tamoxifen, efavirenz, propofol, methadone, and bupropion)
* Have received a hematopoietic stem cell transplant
* Have a second primary malignancy that in the judgment of the investigator and sponsor, may affect the interpretation of the results
* Have an active fungal, bacterial, and/or known viral infection including human immunodeficiency virus (HIV) or viral (A, B, or C) hepatitis (screening is not required)
* Have a history of congestive heart failure with New York Heart Association (NYHA) Class greater than 2 (NYHA Class 1 and 2 are eligible), unstable angina, recent myocardial infarction (within 6 months prior to administration of study drug), or documented history of ventricular arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-06-11 (Actual); Primary Completion 2015-06-26 (Actual); Study Completion 2017-02-24 (Actual)

PRIMARY OUTCOMES:
Number of participants with LY2784544 dose limiting toxicities (DLT) | Baseline through Cycle 1 in Part A (28 day cycles)
Recommended dose range and regimen for Phase 2 studies | Baseline through Cycle 1 in Part B (28 day cycles)

SECONDARY OUTCOMES:
Pharmacokinetics of LY2784544: Maximum concentration (Cmax) | Cycle 1 in Part A and Part B (28 day cycles)
Pharmacokinetics of LY2784544: Area under the concentration-time curve (AUC) | Cycle 1 in Part A and Part B (28 day cycles)
International Working Group (IWG) response | Baseline through last Cycle in Part A and Part B (28 day cycles)
Dynamic International Prognostic Scoring System (DIPSS) Plus | Baseline through last Cycle in Part A and Part B (28 day cycles)
Change in symptom burden as assessed by the Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF) | Baseline, Last Cycle in Part A and Part B
Change in Myeloproliferative Neoplasm (MPN) Physician Symptom Assessment | Baseline, Last Cycle in Part A and Part B

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (9):
- United States (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scottsdale, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fayetteville, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Washington D.C., District of Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Honolulu, Hawaii
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charleston, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milwaukee, Wisconsin